CLINICAL TRIAL: NCT05053867
Title: A Randomized Controlled Trial of Inhaled Tranexamic Acid for the Treatment of Pulmonary Hemorrhage in Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0991; NCI-2021-09676 (Other: NCI-CTRP Clinical Trials Gov Registry)
Record Dates: First submitted 2021-09-02; First posted 2021-09-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hemorrhage; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Inhaled tranexamic acid (Experimental): will receive 500 mg/5ml nebulized tranexamic acid every 8 hours for at least 3 days, and up to 5 days
  Interventions: Drug: tranexamic acid
- Group B: Usual Care (Other): usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: tranexamic acid — Inhaled
  Arms: Group A: Inhaled tranexamic acid
Other: Usual Care — Standard of Care
  Arms: Group B: Usual Care

SUMMARY:
This is a drug study that will examine if inhaled tranexamic acid can improve mortality in patients with cancer-related pulmonary hemorrhage and respiratory failure as compared to usual care.

DETAILED DESCRIPTION:
Primary Objective: To assess the benefit of using nebulized tranexamic acid versus the standard of care on 30 day mortality.

Secondary Objectives: To assess the following outcomes when using nebulized tranexamic acid versus the standard of care:

1. 100 day, ICU and hospital mortality rate
2. Ventilator days at day 30
3. ICU and Hospital Length of Stay
4. PaO2:FIO2 ratio (or SpO2:FIO2 ratio) changes over the first 14 days
5. Time to resolution of pulmonary hemorrhage
6. Rate of recurrence of pulmonary hemorrhage
7. Rate of invasive procedures required to control pulmonary hemorrhage

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Have a diagnosed hematological malignancy
3. Are actively receiving mechanical ventilation
4. Have evidence of pulmonary hemorrhage as defined by either

   1. Persistently bloody secretions upon endotracheal tube suctioning, or
   2. Evidence of diffuse alveolar hemorrhage by bronchoscopic examination
5. Signed informed consent by patient or if the subject lacks decision-making capacity, the subject's legally authorized representative

2.3.2 Exclusion Criteria

Patients excluded from participation in the study if any of the following criteria are met:

1. Presence of a Do Not Resuscitate (DNR), no escalation of care or comfort care order at the time of screening
2. Expected survival < 48 hours
3. Evidence of nasal or oral spillage likely to be the cause of bloody secretions
4. Patients requiring 100% FIO2
5. Known hypersensitivity to tranexamic acid
6. Treatment with inhaled tranexamic acid prior to screening
7. Acquired defective color vision
8. Subarachnoid hemorrhage
9. Deep Venous or arterial thrombus diagnosed within the previous 3 months
10. Seizure disorder on active anti-epileptic therapies
11. Hypersensitivity to tranexamic acid or any of the ingredients
12. Pregnant women will not be eligible and have a negative pregnancy test prior to entering study
13. Patient receiving concurrent anti-fibrinolytic therapy
14. Confirmed active COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
28 day all-cause mortality rate | up to 28 days
  Number of patients who are alive at 28 days following randomization. The difference between 28-day mortality rates between treatment arms will be computed along with a 95% confidence interval (CI) using the approximate standard error reported in Fleiss (1981). Logistic regression will be used to estimate the association between 28-day mortality and study covariates of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Rathi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org